CLINICAL TRIAL: NCT07235124
Title: Psychobiological Correlates of Achievement Motivation and Neurotransmitter Responses to Exercise in Elite Rowers
Brief Title: Motivation and Neurotransmitters in Rowers
Status: Completed | Type: Observational
Sponsor: Poznan University of Physical Education (Other)
Responsible Party: Sponsor
Other Study IDs: LMI60002023
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Healthy
Keywords: Elite athletes; Fatigue; Recovery; Neurotransmitters; Achievement motivation
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Rowers: The study includes 24 national-level male rowers. All participants are healthy, highly trained athletes with at least 3 years of systematic rowing experience and regular intensive training.
  Interventions: Other: 6000-meter rowing ergometer test

INTERVENTIONS:
Other: 6000-meter rowing ergometer test — Participants perform a 6000-meter rowing test on an indoor ergometer at maximal effort to simulate race conditions and induce physiological fatigue.

SUMMARY:
The goal of this observational study is to learn how motivation and body chemistry are linked during and after intense exercise in national-level rowers.

The main questions this study aims to answer are:

Do athletes with higher motivation show different changes in brain chemicals after exercise? How do hormone and neurotransmitter levels change during recovery after exercise?

Participants will:

Complete a motivation questionnaire called the Inventory of Achievement Motivation (LMI) before the exercise test.

Perform a 6000-meter rowing test on an indoor rowing machine. Have blood samples taken three times: before exercise, immediately after exercise, and 1 hour after exercise.

Researchers will measure blood levels of testosterone, cortisol, serotonin, dopamine, beta-endorphin, anandamide (AEA), and 2-arachidonoylglycerol (2-AG).

This study will help researchers understand how motivation and body chemistry work together to influence performance and recovery in highly trained athletes.

DETAILED DESCRIPTION:
This study explores how motivation and body chemistry are connected during and after intense physical exercise in national-level rowers. Researchers want to understand how psychological factors, such as motivation to achieve goals, relate to changes in hormones and brain chemicals that occur with exercise and recovery.

Before the exercise test, participants will complete a motivation questionnaire called the Inventory of Achievement Motivation (LMI). This questionnaire helps identify how strongly a person is driven to perform, overcome challenges, and reach success.

After the questionnaire, each participant will complete a 6000-meter rowing test on an indoor rowing machine. This test is designed to produce a high level of physical effort similar to competition conditions. Blood samples will be taken three times: before the test, immediately after the test, and one hour after recovery.

The blood samples will be used to measure levels of several hormones and neurotransmitters, including testosterone, cortisol, serotonin, dopamine, beta-endorphin, anandamide (AEA), and 2-arachidonoylglycerol (2-AG). These substances are involved in stress response, motivation, reward, and recovery.

Researchers will compare the results from the motivation questionnaire with changes in hormone and neurotransmitter levels. The goal is to find out whether more motivated athletes show different chemical responses to exercise and recovery.

Findings from this study may improve understanding of how the mind and body interact during intense training. This knowledge could help athletes and coaches develop better ways to support motivation, performance, and recovery in high-level sports.

ELIGIBILITY:
Inclusion Criteria:

National-level male rowers Age between 18 and 35 years Minimum of 3 years of systematic rowing training Regular training load (at least 10 sessions per week during the competitive season) Good general health and medical clearance for maximal exercise testing

Exclusion Criteria:

Current illness, injury, or infection Use of medications or dietary supplements that could affect hormone or neurotransmitter levels Smoking or use of psychoactive substances Inadequate sleep or food intake before testing Refusal or inability to provide informed consent

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All participants were recruited and tested at the Central Sports Centre - Olympic Preparation Center (COS OPO) in Wałcz, Poland, during a national team training camp under standardized conditions.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2023-12-02 (Actual)

PRIMARY OUTCOMES:
Changes in serum Cortisol levels | Before exercise, immediately after, and 1 hour after recovery
  Measurement of Cortisol serum concentrations (ng/mL).
Changes in serum Testosterone levels | Before exercise, immediately after, and 1 hour after recovery
  Measurement of Testosterone serum concentrations (ng/mL).
Changes in serum Dopamin levels | Before exercise, immediately after, and 1 hour after recovery
  Measurement of Dopamin serum concentrations (ng/mL).
Changes in serum Serotonin levels | Before exercise, immediately after, and 1 hour after recovery
  Measurement of Serotonin serum concentrations (ng/mL).
Changes in serum Beta-endorphin levels | Before exercise, immediately after, and 1 hour after recovery
  Measurement of Beta-endorphin serum concentrations (ng/mL).
Changes in serum anandamide (AEA) levels | Before exercise, immediately after, and 1 hour after recovery
  Measurement of anandamide (AEA) serum concentrations (ng/mL).
Changes in serum 2-arachidonoylglycerol (2-AG)) levels | Before exercise, immediately after, and 1 hour after recovery
  Measurement of 2-arachidonoylglycerol (2-AG) serum concentrations (ng/mL).

SECONDARY OUTCOMES:
Changes in Testosterone-to-cortisol ratio (T:C) | Before exercise, immediately after, and 1 hour after recovery
  Ratio calculated from serum testosterone and cortisol concentrations (ng/mL), used as an indicator of anabolic-catabolic balance.
Changes in TSerotonin-to-dopamine ratio (S:D) | Before exercise, immediately after, and 1 hour after recovery
  Ratio of serum serotonin to dopamine concentrations (ng/mL), reflecting neurochemical balance related to motivation and fatigue.
Achievement Motivation (LMI score) | Before exercise (baseline)
  Assessment of achievement motivation using the Inventory of Achievement Motivation (LMI). The questionnaire evaluates multiple dimensions of motivation, such as persistence, confidence in success, goal setting, and compensatory effort. Total and subscale scores are analyzed to identify individual motivational profiles.

CONTACTS AND LOCATIONS:
Locations (1):
- Poznań University of Physical Education, Poznan, Greater Poland Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. Data will be used only for internal analysis and dissemination in scientific publications in aggregate form, in accordance with ethical approval.